CLINICAL TRIAL: NCT02447081
Title: Amplatzer™Amulet™ Observational Post-Market Study
Brief Title: Amplatzer™Amulet™ Post-Market Study (Amulet™PMS)
Acronym: Amulet™PMS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10053
Record Dates: First submitted 2015-04-27; First posted 2015-05-18 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation; Thromboembolism; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects implanted with Amulet Device: All subjects who receive the Amulet device will be followed.
  Interventions: Device: Subjects implanted with Amulet Device

INTERVENTIONS:
Device: Subjects implanted with Amulet Device — Percutaneous Left Atrial Appendage occlusion with successful implant of occlusion device.

SUMMARY:
This was a prospective, multicenter, observational, nonrandomized study to compile real world outcome data on the use of the Amulet™ device in non-valvular atrial fibrillation (NVAF) subjects. The study was designed to follow the Instructions For Use (IFU) to gather data on the implant procedure through two years of follow up with the Amulet™ device in a commercial clinical setting."

DETAILED DESCRIPTION:
A total of 1088 subjects were enrolled in the study at 61 sites internationally, outside the United States.

The study assessed acute and late serious adverse events and reports the rate of stroke and bleeding events through 2 years. No formal hypothesis were tested for this observational post-market study.

Each patient was followed at study visits at baseline, implant, 1-3 months, 6 months, 12 months, and 24 months post implant."

ELIGIBILITY:
Inclusion Criteria:

1. Subject with history of paroxysmal, persistent or permanent NVAF
2. Subject who is 18 years or older, or of legal age to give informed consent specific to state and national law
3. Subject who is eligible for an Amulet LAA Occluder device according to current international guidelines and per physician discretion
4. Subject who is willing and capable of providing informed consent, participating in all associated study activities

Exclusion Criteria:

1. Subject with evidence of an intracardiac thrombus
2. Subject with active infection or active endocarditis or other infections producing bacteremia
3. Subject where the placement of the device would interfere with any intracardiac or intravascular structures
4. Subject with any medical disorder that would interfere with completion or evaluation of clinical study results
5. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment per physician discretion)
6. Subject with LAA anatomy that does not accommodate a device per the sizing guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1088 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hildick-Smith, MD, Principal Investigator — Brighton and Sussex University Hospitals; Claudio Tondo, MD PhD, Principal Investigator — University of Milan
Locations (51):
- Fiona Stanley Hospital, Murdoch, Western Australia, Australia
- Universitaire Ziekenhuizen Gasthuisberg, Leuven, Belgium
- Hospital Clinico San Borja Arriaran, Santiago, Chile
- Rigshospitalet, Copenhagen, Denmark
- Finland (2):
  - Helsinki University Central Hospital, Helsinki, Uusimaa
  - Turku University Hospital, Turku
- France (4):
  - Hopital Haut Leveque, Pessac, Aquitaine
  - CHU du Bocage, Dijon, Burgundy
  - CHRU Lille, Lille, North-Calais
  - CHU d'Amiens, Amiens, Picardy
- Germany (17):
  - Klinikum Coburg, Coburg, Bavaria
  - Internistische Klinik Dr. Müller, München-Thalkirchen, Munich, Bavaria
  - Universitaetsklinikum Ulm, Ulm, Bavaria
  - Zentrum fur Herzgesundheit/Kardiologie am Alice Hospital Darmstadt, Darmstadt, Hesse
  - CardioVaskuläres Centrum St. Katharinen, Frankfurt am Main, Hesse
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphal
  - Zentralklinik Bad Berka Gmbh, Bad Berka, Thuringia
  - Zentralklinik Bad Berka, Bad Berka
  - Segeberger Kliniken Gmbh, Bad Segeberg
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Charité - Universitätsmedizin Berlin (CBF), Berlin
  - St. Marien Hospital Bonn, Bonn
  - Herzzentrum Dresden, Dresden
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Klinikum Frankfurt Höchst, Frankfurt
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Rems-Murr-Klinikum Winnenden, Winnenden
- Mater Hospital, Dublin, Ireland
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (8):
  - Nuovo Ospedale Civile Sant'Agostino Estense, Baggiovara, Modena
  - Ospedale dell'Angelo and Ospedale SS Giovanni e Paolo Venezia, Mestre, Veneto
  - Università degli Studi di Padova, Padua, Veneto
  - Azienda Ospedaliera S. Anna e S. Sebastiano, Caserta
  - Ospedale del Cuoro Fondazione C. N. R. Regione Toscana G. Monasterio, Massa
  - Cardiac Arrhythmia Research Center, Centro Cardiologico Monzino, Unveristiy of Milan, Milan
  - San Raffaele Hospital, Milan
  - Ospedale Luigi Sacco, Milan
- Amsterdam Academic Medical Centre, Veenendaal, Netherlands
- Ulleval Universitetssykehus, Oslo, Norway
- Poland (2):
  - Slaskie Centrum Chorob Serca, Warsaw
  - The Cardinal Stefan Wyszynski Institute of Cardiology, Warsaw
- Spain (6):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Island
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital de la Santa Creu I Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Infanta Cristina, Badajoz, Extremadura
  - Hospital Clinic I Provincial de Barcelona, Barcelona
- Karolinska University Hospital Huddinge, Stockholm, Sweden
- United Kingdom (3):
  - Liverpool Heart and Chest Hospital, Liverpool, Northwest England
  - The Royal Sussex Country Hospital, Brighton, South East England
  - St Thomas Hospital, London

REFERENCES:
- [Derived] De Caterina AR, Nielsen-Kudsk JE, Schmidt B, Mazzone P, Fischer S, Lund J, Montorfano M, Gage R, Lam SCC, Berti S. Gender difference in left atrial appendage occlusion outcomes: Results from the Amplatzer Amulet Observational Study. Int J Cardiol Heart Vasc. 2021 Jul 26;35:100848. doi: 10.1016/j.ijcha.2021.100848. eCollection 2021 Aug. PMID 34381870
- [Derived] Piayda K, Hellhammer K, Nielsen-Kudsk JE, Schmidt B, Mazzone P, Berti S, Fischer S, Lund J, Montorfano M, Della Bella P, Gage R, Zeus T. Clinical outcomes of patients undergoing percutaneous left atrial appendage occlusion in general anaesthesia or conscious sedation: data from the prospective global Amplatzer Amulet Occluder Observational Study. BMJ Open. 2021 Mar 24;11(3):e040455. doi: 10.1136/bmjopen-2020-040455. PMID 33762228
- [Derived] Aminian A, De Backer O, Nielsen-Kudsk JE, Mazzone P, Berti S, Fischer S, Lund J, Montorfano M, Lam SCC, Freixa X, Gage R, Diener HC, Schmidt B. Incidence and clinical impact of major bleeding following left atrial appendage occlusion: insights from the Amplatzer Amulet Observational Post-Market Study. EuroIntervention. 2021 Oct 20;17(9):774-782. doi: 10.4244/EIJ-D-20-01309. PMID 33495144
- [Derived] Tarantini G, D'Amico G, Schmidt B, Mazzone P, Berti S, Fischer S, Lund J, Montorfano M, Della Bella P, Lam SCC, Cruz-Gonzalez I, Gage R, Zhao H, Omran H, Odenstedt J, Nielsen-Kudsk JE. The Impact of CHA2DS2-VASc and HAS-BLED Scores on Clinical Outcomes in the Amplatzer Amulet Study. JACC Cardiovasc Interv. 2020 Sep 28;13(18):2099-2108. doi: 10.1016/j.jcin.2020.06.003. PMID 32972570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1088 subjects were enrolled and attempted implant with Amulet left atrial appendage occluder conducted at 61 sites between June 01, 2015 and September 19, 2016. The final study visit at 2 years post-implant was completed by 864 subjects, with the last study visit occurring in October 2018.
Period: Overall Study
Arm/Group | Subjects Implanted With Amulet Device
Started | 1088
Completed | 864
Not Completed | 224
Not completed — Death | 161
Not completed — Lost to Follow-up | 36
Not completed — Visit not completed | 17
Not completed — unsuccessful implant procedure | 10

BASELINE CHARACTERISTICS:
Groups:
- Subjects Implanted With Amulet Device: All subjects who received the Amulet device were followed.
  Subjects implanted with Amulet Device: Percutaneous Left Atrial Appendage occlusion with successful implant of occlusion device.
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1088
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 122
  >=65 years | 966
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 386
  Male | 702
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 59
  Spain | 105
  Netherlands | 1
  Sweden | 13
  Belgium | 17
  Norway | 5
  Finland | 55
  Poland | 26
  Denmark | 62
  Italy | 178
  Israel | 1
  Australia | 70
  France | 65
  Chile | 6
  Germany | 378
  Hong Kong | 41
  Switzerland | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Serious Adverse Events
Description: Acute adverse events were defined as those serious events with an onset date ≤ 7 days post-procedure
Time Frame: 0 to 7 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1088
Participants | 83

2. Primary Outcome: Number of Participants With Late Serious Adverse Events Greater Than 7 Days Post Procedure
Description: Late adverse events were defined as those serious events with an onset date > 7 days post-procedure
Time Frame: 7 days through 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1088
Participants | 504

3. Primary Outcome: Number of Participants With Ischemic Stroke, Systemic Embolism and Cardiovascular Death
Description: Occurrence of ischemic stroke, systemic embolism, and cardiovascular death through 2 years
Time Frame: Implant through 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1088
Participants | 122

4. Primary Outcome: Number of Participants With Major Bleeding Events
Description: Clinical events were adjudicated by the CEC as major bleeding events if they met the definition of Type 3 or greater on the Bleeding Academic Research Consortium (BARC) scale.
Time Frame: Implant through 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1088
Participants | 110

5. Secondary Outcome: Number of Participants With Technical Success
Description: Technical success is defined as successful implantation of the Amulet device in the left arterial appendage (LAA).
Time Frame: During implant procedure, approximately 30 to 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1088
Participants | 1078

6. Secondary Outcome: Number of Participants With Procedural Success
Description: Procedural success is based on Amulet device being implanted day 0 through hospital discharge, on average one night stay (day 1). Amulet device implanted and subject discharged the following day without an adverse event
Time Frame: During the implant procedure and hospital stay, approximately 1 or 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1088
Participants | 1039

7. Secondary Outcome: Number of Participants With Oral Anti-coagulation Usage
Time Frame: At discharge, approximately 1 or 2 days after the procedure
Population: The number of participates completing a study visit at the Time Frame
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1074
Participants
  OAC without anti-platelet therapy | 49
  OAC with antiplatelet therapy | 71

8. Secondary Outcome: Number of Participants With Oral Anti-coagulation Usage
Time Frame: At 1 to 3 months
Population: The number of participates completing a study visit at the Time Frame
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1018
Participants
  OAC without anti-platelet therapy | 29
  OAC with anti-platelet therapy | 34

9. Secondary Outcome: Number of Participants With Oral Anti-coagulation Usage
Time Frame: At 6 months
Population: The number of participates completing a study visit at the Time Frame
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 1009
Participants
  OAC without anti-platelet therapy | 33
  OAC with anti-platelet therapy | 23

10. Secondary Outcome: Number of Participants With Oral Anti-coagulation Usage
Time Frame: At 12 months
Population: The number of participates completing a study visit at the Time Frame
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 950
Participants
  OAC without anti-platelet therapy | 35
  OAC with anti-platelet therapy | 21

11. Secondary Outcome: Number of Participants With Oral Anti-coagulation Usage
Time Frame: At 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted With Amulet Device
Number analyzed (Participants) | 864
Participants
  OAC without anti-platelet therapy | 38
  OAC with anti-platelet therapy | 19

ADVERSE EVENTS:
Time Frame: 2 years
Description: Non-serious adverse event information was not analyzed.
Arm/Group | Subjects Implanted With Amulet Device
All-Cause Mortality (participants affected / at risk) | 161/1088
Serious Adverse Events (participants affected / at risk) | 538/1088
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Implanted With Amulet Device (N=1088)
Abdominal Pain (Gastrointestinal disorders) | 2
Acute bacterial endocarditis (Cardiac disorders) | 1
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 5
Acute erosive gastritis (Gastrointestinal disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Acute pancreatitis (Gastrointestinal disorders) | 1
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Acute renal failure (Renal and urinary disorders) | 20
Acute subdural hematoma (Nervous system disorders) | 1
Adult respiratory distress syndrome(ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Air embolus (Respiratory, thoracic and mediastinal disorders) | 1
Alcohol intoxication (Injury, poisoning and procedural complications) | 2
Anemias (Blood and lymphatic system disorders) | 26
Angina pectoris (Cardiac disorders) | 8
Aortic dissection (Cardiac disorders) | 2
Aortic value stenosis (Cardiac disorders) | 5
Aphasia (Nervous system disorders) | 1
Arm fracture (Musculoskeletal and connective tissue disorders) | 2
Arterial hypertension/Hypertension (Cardiac disorders) | 5
Ascites (Cardiac disorders) | 7
Aspiration Pneumonia/Necrotizing pneumonia/Aspiration of vomitus (Gastrointestinal disorders) | 4
Atrial fibrillation (Cardiac disorders) | 37
Atrial flutter (Cardiac disorders) | 8
Atrial tachycardia (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 5
Atrioventricular dissociation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bacterial infection (Infections and infestations) | 19
Bacterial infections of the skin (Infections and infestations) | 7
Benign Tumors (Gastrointestinal disorders) | 2
Bleeding (Blood and lymphatic system disorders) | 6
Bowel Obstruction (Gastrointestinal disorders) | 2
Brain Tumor (Nervous system disorders) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Burns (Injury, poisoning and procedural complications) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23
Cardiac Arrest (Cardiac disorders) | 12
Cardiac Decompensation (Cardiac disorders) | 15
Cardiac Perforation (Cardiac disorders) | 1
Cardiogenic Shock (Cardiac disorders) | 1
Cellulitis (Infections and infestations) | 2
Cerebral Aneurysm (Nervous system disorders) | 1
Chest Pain (Cardiac disorders) | 7
Cholecystitis (Hepatobiliary disorders) | 2
Choledocholithiaisis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 4
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 2
Chronic Renal Failure (General disorders) | 6
Chronic Subdural Hematoma (Nervous system disorders) | 1
Clostridum difficile Infection (Infections and infestations) | 4
Cognitive Impairment (Psychiatric disorders) | 1
Colitis (Gastrointestinal disorders) | 4
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Compression Fracture (Injury, poisoning and procedural complications) | 2
Confusion (General disorders) | 4
Congestive Heart Failure (Cardiac disorders) | 13
Constipation (Gastrointestinal disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 2
Cutaneous Abcesses (Skin and subcutaneous tissue disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Decompensated Heart Failure (Cardiac disorders) | 62
Deep Vein/Venous Thrombosis (Vascular disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Delirium (Psychiatric disorders) | 4
Dementia (Nervous system disorders) | 1
Device Embolization (Surgical and medical procedures) | 2
Diabetes Mellitus (Endocrine disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Diverticulitis (Gastrointestinal disorders) | 1
Diverticulosis (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Drug Side Effect (General disorders) | 1
Duodenal Ulcer (Gastrointestinal disorders) | 2
Dyspnea (Cardiac disorders) | 2
EKG Abnormalities (Cardiac disorders) | 1
Elective Cardiac Surgery (Surgical and medical procedures) | 1
Emesis/Vomiting (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Epididymitis (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Eye Bleed (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 9
Fever (Injury, poisoning and procedural complications) | 4
Fracture (Musculoskeletal and connective tissue disorders) | 6
Fungal Skin Infection (Infections and infestations) | 1
Gastritis (Gastrointestinal disorders) | 4
Gastroenteritis (Gastrointestinal disorders) | 4
Gastrointestinal Bleeding (Gastrointestinal disorders) | 57
Gastroparesis (Gastrointestinal disorders) | 1
Generalized Seizures (Nervous system disorders) | 1
Glaucoma (Eye disorders) | 1
Gout (General disorders) | 4
Hallucinations (Psychiatric disorders) | 1
Heart Block (Cardiac disorders) | 1
Heart Failure (Cardiac disorders) | 6
Heartburn (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 2
Hematoma (Vascular disorders) | 5
Hematuria (Renal and urinary disorders) | 12
Hemiblock (Fascicular Block) (Cardiac disorders) | 1
Hemoperitoneum (Gastrointestinal disorders) | 1
Hemoptysis (General disorders) | 2
Hepatic and Biliary Disorders (Hepatobiliary disorders) | 1
Hernia (Congenital, familial and genetic disorders) | 1
Hip Dislocation (Musculoskeletal and connective tissue disorders) | 1
Hip Fracture (Musculoskeletal and connective tissue disorders) | 7
Hip Pain (Musculoskeletal and connective tissue disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertensive Crisis (Vascular disorders) | 4
Hyperthyroidism (Endocrine disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (General disorders) | 1
Hypotension (Cardiac disorders) | 5
Hypothermia (General disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Infective/Bacterial Endocarditis (Infections and infestations) | 1
Inguinal Hernia (Gastrointestinal disorders) | 2
Intracerebral Haemorrhage (Nervous system disorders) | 10
Iron-Deficiency Anemia (Gastrointestinal disorders) | 3
Ischemic Stroke (Cardiac disorders) | 39
Knee Pain (Musculoskeletal and connective tissue disorders) | 1
Leukemias (Blood and lymphatic system disorders) | 2
Low Back Pain (Musculoskeletal and connective tissue disorders) | 3
Lumbar Spondylosis (Musculoskeletal and connective tissue disorders) | 1
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melena (Blood and lymphatic system disorders) | 2
Miscellaneous Infections (Infections and infestations) | 1
Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 5
Multiple Organ Failure (General disorders) | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3
Myocardial Infarction (Cardiac disorders) | 10
Nephrolithiasis (Renal and urinary disorders) | 2
Neurological Hematoma (Nervous system disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 2
Ocular Hemorrhage (Eye disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 1
Osler Weber Rendu Syndrome (Congenital, familial and genetic disorders) | 1
Osteoarthritis/Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 2
Overdose (Cardiac disorders) | 1
Pain (General disorders) | 2
Palpitations (Cardiac disorders) | 1
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Parkinson's Disease (Nervous system disorders) | 1
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1
Perforated Appendix (Gastrointestinal disorders) | 1
Pericardial Effusion (Cardiac disorders) | 9
Pericardial Tamponade (Cardiac disorders) | 11
Peripheral Arterial Occlusion (Cardiac disorders) | 6
Peripheral Vascular Disease (Cardiac disorders) | 7
Persistent Atrial Fibrillation (Cardiac disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 33
Pneumonia Caused By Gram-Negative Bacilli (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia in the Compromised Host (Respiratory, thoracic and mediastinal disorders) | 2
Polyneuropathy (Nervous system disorders) | 1
Portal-Systemic Encephalopathy (Nervous system disorders) | 1
Pressure Sores (Skin and subcutaneous tissue disorders) | 1
Presyncope (General disorders) | 3
Primary Biliary Cirrhosis (Hepatobiliary disorders) | 2
Psychogenic Event (Psychiatric disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Vascular disorders) | 2
Raynaud's Syndrome (Vascular disorders) | 2
Renal Failure (General disorders) | 9
Renal Insufficiency (Renal and urinary disorders) | 2
Respiratory Failure (Injury, poisoning and procedural complications) | 1
Rheumotologic Disease (Musculoskeletal and connective tissue disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 1
Second Degree Heart Block (Cardiac disorders) | 1
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 14
Sepsis (Infections and infestations) | 19
Septicemia (Infections and infestations) | 2
Shock (General disorders) | 3
Sick Sinus Syndrome (Cardiac disorders) | 2
Simple Partial Seizures (Nervous system disorders) | 1
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 3
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Status Epilepticus (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Subdural Haemorrhage (Nervous system disorders) | 1
Suicide Attempt (Psychiatric disorders) | 1
Sustained Atrial Fibrillation (Cardiac disorders) | 1
Syncope (General disorders) | 11
TEE-Related Event (Cardiac disorders) | 1
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 1
Thrombus (Cardiac disorders) | 1
Thrombus on Device (Cardiac disorders) | 19
Torsade de Pointes (Cardiac disorders) | 1
Transient Ischemic Attack (TIA) (General disorders) | 14
Trauma (General disorders) | 9
Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation Valve (Cardiac disorders) | 1
Unstable Angina (Cardiac disorders) | 7
Unsustained/Nonsustained Ventricular Tachy/Cardiac Arrhythmia (Cardiac disorders) | 1
Urethral Dysfunction (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 7
Urinary Tract Infections (Renal and urinary disorders) | 11
VASC AV Fistula (Surgical and medical procedures) | 4
VASC Bleeding (Vascular disorders) | 4
VASC Hematoma (Vascular disorders) | 4
VASC Pseudoaneurysm (Injury, poisoning and procedural complications) | 4
Vascular Dissection (Cardiac disorders) | 1
Vascular Ischemia (Cardiac disorders) | 3
Vaso Vagal Response (Nervous system disorders) | 1
Ventricular Fibrillation (Cardiac disorders) | 3
Ventricular Tachycardia (Cardiac disorders) | 4
Vessel Occlusion (Vascular disorders) | 1
Viral Syndrome (Infections and infestations) | 1
Weakness (General disorders) | 1
Wound Dehiscence (General disorders) | 1
Other (General disorders) | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02447081/Prot_SAP_000.pdf